CLINICAL TRIAL: NCT04467788
Title: Effectiveness of Computer-Aided Versus Clinical Simulation Sessions on Knowledge, Attitude and Practice of Ergonomics Among A Group of Dental Interns: A Randomized Controlled Trial
Brief Title: Effectiveness of Computer-Aided Versus Clinical Simulation Sessions on Knowledge, Attitude and Practice of Ergonomics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Saad Mohamed Ali, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NSaad
Record Dates: First submitted 2020-06-29; First posted 2020-07-13 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Occupational Problems
Keywords: Ergonomics in dentistry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-aided session (Active Comparator): Training on ergonomic principles in dentistry will be given to the participants through Computer-Aided sessions, including explaining videos on proper postures in dental practice .
  Interventions: Other: Computer-aided sessions
- Clinical Simulation Session (Active Comparator): Training on ergonomic principles in dentistry will be given to the participants through clinical simulation sessions showing the proper postures in dental practice.
  Interventions: Other: Clinical simulation sessions

INTERVENTIONS:
Other: Computer-aided sessions — Changing participants' KAP of ergonomics in dentistry
  Arms: Computer-aided session
Other: Clinical simulation sessions — Changing participants' KAP of ergonomics in dentistry
  Arms: Clinical Simulation Session

SUMMARY:
A healthy dentist is one of the most important components of a successful dental practice. It is estimated that more than half of practitioners have some kind of painful work-related musculoskeletal disorders.

It was reported that 80% of dental students were not aware of ergonomic posture during dental procedures. It is believed that dental students with knowledge of ergonomic principals would be able to maintain their health. Some studies demonstrated that the frequency and severity of WMSDs might decrease by training the dentists on ergonomic principles.

DETAILED DESCRIPTION:
This study will be carried out on dental interns in Department of Pediatric Dentistry and Dental Public Health, in Faculty of Dentistry-Cairo University. The procedures will be carried out by postgraduate student Nourhan Saad Mohamed who has M.D.S. (2018) - Cairo University- Egypt, and works as Assistant Lecturer in Future University in Egypt. The procedures will be done without assistant at a lecture room and outpatient clinic of Pediatric Dentistry in Cairo University.

At baseline, evaluation of knowledge, attitude and practice (KAP) on ergonomics in dentistry will be do e through a self-structured questionnaire.

Afterwards, the participants will be split into two groups. One group will recieve training on ergonomic principles through clinical simulation session, while the other group will recieve training through Computer-aided sessions.

KAP will be re-evaluated after the training sessions to evaluate the change in KAP about ergonomics.

ELIGIBILITY:
Inclusion Criteria:

* Dental interns who accept to participate in the study.
* Graduates of governmental or private dental schools.

Exclusion Criteria:

* Interns with history of chronic musculoskeletal disorders.
* Interns who perform other physical activities which required forced posture.
* Interns with history of fracture in the ribs or vertebrae.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
KAP questionnaire on ergonomics in dentistry | 1 questionnaire for 15 minutes before the learning modules
  At baseline, assessment of the knowledge, attitude and practice of dental interns regarding ergonomics in Dentistry will be done before the educational module assigned to each group. The questionnaire will include 25 multiple choice questions, each question will score 4 with the total questionnaire out of 100.
  The questionnaire that will score 75 or less will considered as failed.

SECONDARY OUTCOMES:
Change in knowledge, attitude & practice of ergonomics after interactive learning about ergonomics in dentistry through computer-aided sessions on ergonomic principles. | 1 questionnaire (15 minutes) after the computer aided session and another questionnaire (15 minutes)at the end of internship round
  Assessment of the knowledge, attitude and practice of dental interns regarding ergonomics in Dentistry will be done after the educational module assigned to the group. The questionnaire will include 25 multiple choice questions, each question will score 4 with the total questionnaire out of 100.
  The questionnaire that will score 75 or less will considered as failed.
Change in knowledge, attitude & practice of ergonomics after interactive learning about ergonomics in dentistry through clinical simulation sessions on ergonomic principles | 1 questionnaire (15 minutes) after the clinical simulation session and another questionnaire (15 minutes)at the end of internship round
  Assessment of the knowledge, attitude and practice of dental interns regarding ergonomics in Dentistry will be done after the educational module assigned to the group. The questionnaire will include 25 multiple choice questions, each question will score 4 with the total questionnaire out of 100.
  The questionnaire that will score 75 or less will considered as failed.